CLINICAL TRIAL: NCT05009225
Title: Reducing Variation in Hospitalization and Processes of Care in Emergency Department Patients With Atrial Fibrillation: A Stepped Wedge Cluster Randomized Trial
Brief Title: Clinical Decision Support for Atrial Fibrillation and Flutter
Status: Active, not recruiting | Type: Observational
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: 1279670
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation and Flutter
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Comprehensive ED AF management tool — Managing atrial fibrillation (AF) patients in the emergency department (ED) is complex, often requiring many separate decisions: How to best reduce the heart rate? Should emergency physicians attempt cardioversion? If so, how? Does this patient need stroke prevention? The investigators' CDSS provides emergency physicians with a one-stop, evidence-based resource that addresses all aspects of ED AF management.

SUMMARY:
Atrial fibrillation (AF) is a major public health problem: it impairs quality of life and independently heightens the risks of ischemic stroke, heart failure and all-cause mortality. AF is a common reason for presenting to emergency departments (ED) in Kaiser Permanente Northern California (KPNC) and is associated with frequent hospitalization. Additionally, inter-facility hospitalization rates for AF vary across KPNC. Improvements in modifiable components of ED AF care could potentially reduce low-yield hospitalizations and the associated costs, patient inconveniences, and complications that can ensue. Real-time clinical decision support systems (CDSS) can transform entrenched physician practices and improve patient outcomes. The investigators will conduct a stepped-wedge cluster randomized trial of a CDSS intervention across 13 KPNC EDs for the comprehensive management of acute AF with the following three aims: 1) To evaluate the impact of the CDSS intervention on index hospitalization rates; 2) To evaluate the impact of the CDSS intervention on ED AF rate and rhythm control process-of-care metrics; and 3) To evaluate the impact of the CDSS intervention on AF stroke prevention actions for eligible participants at the time of ED discharge. The investigators hypothesize that the CDSS intervention will safely reduce index hospitalization rates, improve rate and rhythm control process-of-care metrics, and increase stroke prevention actions for eligible participants at ED discharge and within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18y) KPNC members presenting to the ED with a primary ED diagnosis of atrial fibrillation/flutter (AF/FL). Subjects who meet criteria will be identified electronically within the CDSS tool in the electronic health record.

Exclusion Criteria:

* Children (<18y).
* Non-members of KPNC.
* Patients who were prisoners, pregnant, receiving hospice or palliative care, or who left against medical advice at the index encounter for AF/FL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to KPNC emergency departments with eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients who were hospitalized | Through emergency department visit, an average of 8 hours
Number of patients who received sustained rate-reduction medications | Through emergency department visit, an average of 8 hours
Number of patients who received stroke prevention interventions | Through emergency department visit, an average of 8 hours

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Kaiser Permanente Antioch Emergency Department, Antioch, California
  - Kaiser Permanente Fremont Emergency Department, Fremont, California
  - Kaiser Permanente Manteca Medical Center, Manteca, California
  - Kaiser Permanente Modesto Medical Center, Modesto, California
  - Kaiser Permanente Oakland Emergency Department, Oakland, California
  - Kaiser Permanente Richmond Emergency Department, Richmond, California
  - Kaiser Permanente Roseville Emergency Department, Roseville, California
  - Kaiser Permanente South Sacramento Emergency Department, Sacramento, California
  - Kaiser Permanente Sacramento Emergency Department, Sacramento, California
  - Kaiser Permanente San Francisco Emergency Department, San Francisco, California
  - Kaiser Permanente San Jose Emergency Department, San Jose, California
  - Kaiser Permanente San Leandro Emergency Department, San Leandro, California
  - Kaiser Permanente San Rafael Emergency Department, San Rafael, California
  - Kaiser Permanente Santa Clara Emergency Department, Santa Clara, California
  - Kaiser Permanente South San Francisco Emergency Department, South San Francisco, California
  - Kaiser Permanente Walnut Creek Medical Center, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vinson DR, Warton EM, Durant EJ, Mark DG, Ballard DW, Hofmann ER, Sax DR, Kene MV, Lin JS, Poth LS, Ghiya MS, Ganapathy A, Whiteley PM, Bouvet SC, Rauchwerger AS, Zhang JY, Shan J, DiLena DD, Kea B, Pai AP, Loyles JB, Solomon MD, Go AS, Reed ME. Decision Support Intervention and Anticoagulation for Emergency Department Atrial Fibrillation: The O'CAFE Stepped-Wedge Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2443097. doi: 10.1001/jamanetworkopen.2024.43097. PMID 39504024
- [Derived] Vinson DR, Rauchwerger AS, Karadi CA, Shan J, Warton EM, Zhang JY, Ballard DW, Mark DG, Hofmann ER, Cotton DM, Durant EJ, Lin JS, Sax DR, Poth LS, Gamboa SH, Ghiya MS, Kene MV, Ganapathy A, Whiteley PM, Bouvet SC, Babakhanian L, Kwok EW, Solomon MD, Go AS, Reed ME; Kaiser Permanente CREST Network. Clinical decision support to Optimize Care of patients with Atrial Fibrillation or flutter in the Emergency department: protocol of a stepped-wedge cluster randomized pragmatic trial (O'CAFE trial). Trials. 2023 Mar 31;24(1):246. doi: 10.1186/s13063-023-07230-2. PMID 37004068